CLINICAL TRIAL: NCT02923167
Title: Robotic-assisted Therapy to Improve Manual Dexterity in Children With Cerebral Palsy: a Pilot Study on Clinical Outcomes and Muscle Synergies as a Possible Predictor of Response
Brief Title: Robotic-assisted Therapy to Improve Manual Dexterity in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, PhD, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000926
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy
Keywords: CP; Cerebral Palsy; Robotic; Hand; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic-assisted training of the hand (Experimental): Training will be performed using the Amadeo®. The computer-controlled device maintains participants' forearm in a secure position using Velcro straps. Each training session will include 30 minutes of active movements that can be divided into up to 3 bouts of 10 minutes depending on participant's fatigue. Training will take place up to 4 times per week for a total of 18 sessions over up to 7 weeks. Sessions will last approximately 60 minutes (including setup, training, and rest between each bout).
  Interventions: Device: Robotic-assisted training of the hand

INTERVENTIONS:
Device: Robotic-assisted training of the hand — Training will be performed using the Amadeo®. The computer-controlled device maintains participants' forearm in a secure position using Velcro straps. Each training session will include 30 minutes of active movements that can be divided into up to 3 bouts of 10 minutes depending on participant's fatigue. Training will take place up to 4 times per week for a total of 18 sessions over up to 7 weeks. Sessions will last approximately 60 minutes (including setup, training, and rest between each bout).
  Other Names: Amadeo® - Tyromotion

SUMMARY:
This is an intervention study including a baseline data collection, 6 weeks of robot-assisted training targeting hand dexterity, and a post-intervention data collection. The study will be conducted in the Motion Analysis Laboratory at Spaulding Rehabilitation Hospital, Boston, MA. This study aims to assess the effectiveness of a robot-assisted training on hand dexterity and quality of life in children with cerebral palsy. Additionally, the investigators will study the relationship between muscle synergies and the outcomes of robot-assisted training.

DETAILED DESCRIPTION:
Participants will be assessed 2 times - before and after training with the robot. All the testing and training will be done at Spaulding Rehabilitation Hospital and will include:

Clinical tests:

* A physical examination during which the investigators will measure range of motion and muscular strength at the shoulder, elbow, forearm, wrist, and fingers.
* A test to assess spasticity at the shoulder, elbow, forearm, and wrist.
* A test to evaluate upper extremity function.
* A test to assess unilateral gross manual dexterity.
* A test to assess quality of life (social wellbeing and acceptance, feelings about functioning, participation and physical health, emotional wellbeing and self-esteem, access to service, pain and impact of disability, and family health).

Muscle activity tests:

• A test to get detailed measures of how well participant can perform movements. The measures collected will include the movements of fingers, hands, and arms while picking up different objects. Movements will be tracked by attaching small reflective markers to the fingers, hands, and arms of the participant. Special cameras will be used to collect data. Special sensors (called electromyographic - EMG - sensors) will be attached to the hands and arms to tell the investigators when and how muscles are recruited to generate the movements.

Training with the Robot:

Study participants will undergo robot-assisted training for 18 times - up to 4 times per week during a period of approximately 7 weeks. The training sessions will be carried out by trained study staff. The robot will assist study participants to perform the movements while they attempt to move their fingers to control computer games. The assistance provided by the robot will be adjusted to the ability of each participant to move their hand. Each training session will last about 1 hour. This will include about 20 minutes of stretching exercises, setup time, and warm-up exercises. Study participants will be encouraged to ask for rest breaks whenever needed. The investigators will closely monitor study participants during all study sessions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy (CP) with upper-limb impairment
* 6 to 18 years of age.
* Manual Ability Classification Scale Level II or III.
* Ability to communicate pain or discomfort.

Exclusion Criteria:

* Use of upper-limb robotics for motor training within the last 3 months.
* Contraindication to robotic-assisted manual training such acute and pronounced pain symptoms despite conventional pain therapy of the upper-limb, lack of compliance, high-grade ataxia, advanced osteoporosis, and fractures of the upper-limb.
* Modified Ashworth Scale (MAS) of 4 in the upper-limb.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spauding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic-assisted Training of the Hand
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Diagnosis [Count of Participants; unit: Participants] — Population: Whereas the primary objective of the study was to assess the effects of robot-assisted training in children with Cerebral Palsy, we requested a protocol exception to evaluate the effects of robot-assisted training in 1 child with stroke.
  Participants
    Diagnosis - Cerebral Palsy: number analyzed (Participants) | 5
    Diagnosis - Cerebral Palsy | 5
    Diagnosis - Stroke: number analyzed (Participants) | 1
    Diagnosis - Stroke | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Upper Extremity Skills Test (QUEST) Score - Section on Dissociated Movements
Description: Upper extremity function assessment (section on dissociated movements). The QUEST is a tool that evaluates the quality of upper extremity function. Data is reported on a scale from 0 to 100 for each assessment. The change from baseline to post-intervention is calculated by taking the difference between the value gathered pre-intervention and the value gathered post-intervention.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: We were unable to collect data from 3 study participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Robotic-assisted Training of the Hand: Training will be performed using the Amadeo®. The computer-controlled device maintains participants' forearm in a secure position using Velcro straps. Each training session will include 30 minutes of active movements that can be divided into up to 3 bouts of 10 minutes depending on participant fatigue. Training will take place up to 4 times per week for a total of 18 sessions over up to 7 weeks. Sessions will last approximately 60 minutes (including setup, training, and rest between each bout).
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 3
units on a scale | 3.5 (4.4)

2. Primary Outcome: Change in Quality of Upper Extremity Skills Test (QUEST) Score - Section on Grasp
Description: Upper extremity function assessment (section on grasp). The QUEST is a tool that evaluates the quality of upper extremity function. Data is reported on a scale from 0 to 100 for each assessment. The change from baseline to post-intervention is calculated by taking the difference between the value gathered pre-intervention and the value gathered post-intervention.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: We were unable to collect data from 3 study participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 3
units on a scale | 12.1 (20.2)

3. Secondary Outcome: Change in Box and Block Test Score
Description: Gross manual dexterity assessment. The test is administered by using a wooden box divided in two compartments. At the beginning of the test, 150 wooden blocks are positioned in one of these compartments. Then study participants are instructed to move, one by one, the maximum number of wooden blocks from one compartment to the other one in a time interval of 1 minute. The result of the test is the number of wooden blocks moved in 1 minute. The change from baseline to post-intervention is calculated by taking the difference between the value gathered pre-intervention and the value gathered post-intervention.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: We were unable to collect data from 3 study participants.
Measure: Mean (Standard Deviation); unit: wooden blocks
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 3
wooden blocks | 1.0 (2.0)

4. Secondary Outcome: Change in Cerebral Palsy Quality of Life Questionnaire Score - Child
Description: Questionnaire for evaluation of quality of life as reported by the child. The questionnaire covers different domains (e.g. social wellbeing and acceptance). Data is reported on a scale from 0 to 100. The change from baseline to post-intervention is calculated by taking the difference between the value gathered pre-intervention and the value gathered post-intervention. The change from baseline to follow-up is calculated by taking the difference between the value gathered pre-intervention and the value gathered at one month follow-up.
Time Frame: Data collected at baseline, at completion of the 7-week intervention, and at one month follow-up
Population: We were unable to collect data from 4 study participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 2
units on a scale
  Baseline vs post-intervention | 1.1 (2.3)
  Baseline vs follow-up assessment | 2.4 (4.1)

5. Secondary Outcome: Change in Number of Muscle Synergies
Description: Subjects will be asked to reach and grasp objects of different sizes and shapes. Surface electromyographic (EMG) activity will be collected from 16 muscles of the upper-limb. EMG data is then analyzed using a mathematical technique (referred to as non-negative matrix factorization) that allows researchers to quantify patterns of co-activation among muscles. The number of muscle synergies necessary to accurately reconstruct the individual EMG channel recordings will be herein considered.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: We were able to collect data of sufficient quality to enable the proposed analyses only for one subject. We observed 5 muscle synergies both at baseline and at completion of the 7-week intervention.
Measure: Number; unit: muscle synergies
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 1
muscle synergies | 0

6. Secondary Outcome: Change in Modified Ashworth Scale Score
Description: Upper extremity muscle spasticity assessment. This scale is administered by manually moving the subject's body segments and evaluate if an involuntary (reflex) response of muscles interfere with the passive movement. If testing a muscle that primarily flexes a joint, the rehabilitation specialist evaluating the subject places the joint in a maximally flexed position and moves it to a position of maximal extension over one second. If testing a muscle that primarily extends a joint, the rehabilitation specialist evaluating the subject places the joint in a maximally extended position and moves to a position of maximal flexion over one second. Spasticity causes a contraction resisting the movement. The strength of the contraction (i.e. force involuntarily generated by muscles) is evaluated on a scale from 0 to 4. The change from baseline to post-intervention is calculated by taking the difference between the value gathered pre-intervention and the value gathered post-intervention.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: We were unable to collect data from 5 study participants.
Measure: Number; unit: units on a scale
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 1
units on a scale | -0.5

7. Secondary Outcome: Change in Cerebral Palsy Quality of Life Questionnaire Score - Caregiver
Description: Questionnaire for evaluation of quality of life as reported by the caregiver. The questionnaire covers different domains (e.g. social wellbeing and acceptance). Data is reported on a scale from 0 to 100. The change from baseline to post-intervention is calculated by taking the difference between the value gathered pre-intervention and the value gathered post-intervention. The change from baseline to follow-up is calculated by taking the difference between the value gathered pre-intervention and the value gathered at one month follow-up.
Time Frame: Data collected at baseline, at completion of the 7-week intervention, and at one month follow-up
Population: We were unable to collect data from 3 study participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 3
units on a scale
  Baseline vs post-intervention | 4.0 (5.1)
  Baseline vs follow-up assessment | 4.0 (4.1)

8. Secondary Outcome: Synergy Similarity
Description: Subjects will be asked to reach and grasp objects of different sizes and shapes. Surface electromyographic (EMG) activity will be collected from 16 muscles of the upper-limb. EMG data is then analyzed using a mathematical technique (referred to as non-negative matrix factorization) that allows researchers to quantify patterns of co-activation among muscles. The similarity among muscle synergies is estimated by computing the scalar product between corresponding muscle synergies. Results are reported individually for each muscle synergy. The minimum scalar product is 0 and it means that the synergies (pre- vs post-interventions) are highly dissimilar. The maximum scalar product is 1 and it means that the synergies (pre- vs post-interventions) are identical.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: as for outcome 5
Measure: Number; unit: units on a scale
Arm/Group | Robotic-assisted Training of the Hand
Number analyzed (Participants) | 1
units on a scale
  Similarity for synergy 1 | 0.87
  Similarity for synergy 2 | 0.94
  Similarity for synergy 3 | 0.96
  Similarity for synergy 4 | 0.77
  Similarity for synergy 5 | 0.83

ADVERSE EVENTS:
Time Frame: During each 1-hour session, for a total of 18 sessions over 7 weeks
Arm/Group | Robotic-assisted Training of the Hand
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic-assisted Training of the Hand (N=6)
Unanticipated adverse event (General disorders) | 1 (1) — Subject feeling unwell

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT02923167/Prot_SAP_001.pdf